CLINICAL TRIAL: NCT03898479
Title: A Multicenter, Open-Label, Extension Study to Assess the Long-Term Safety and Efficacy of CTP-543 in Adult Patients With Moderate to Severe Alopecia Areata
Brief Title: Extension Study to Evaluate Safety and Efficacy of CTP-543 in Adults With Alopecia Areata
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Organization: Sun Pharmaceutical Industries Limited (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP543.5001
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTP-543 (Experimental): Patients who previously completed a qualifying CTP-543 clinical trial
  Interventions: Drug: CTP-543

INTERVENTIONS:
Drug: CTP-543 — Twice daily dosing

SUMMARY:
The overall objectives of the study are to evaluate long-term safety of CTP-543 and to assess long-term effects of CTP-543 on treating hair loss in adult patients with chronic, moderate to severe alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* Have completed 24 weeks of treatment in a previous qualifying CTP-543 clinical trial

Exclusion Criteria:

* Active scalp inflammation, psoriasis, or seborrheic dermatitis requiring topical treatment to the scalp, significant trauma to the scalp, or untreated actinic keratosis
* Females who are nursing, pregnant, or planning to become pregnant while in the study, and for 30 days after last dose of study medication
* Donation of blood at any point throughout the study and for 30 days after last dose of study medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-04-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 332 weeks
Effect of CTP-543 on treating hair loss as measured by the Severity of Alopecia Tool (SALT) | 332 weeks

CONTACTS AND LOCATIONS:
Locations (91):
- United States (72):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - Alliance Dermatology & MOHS Center, Phoenix, Arizona
  - Center for Dermatology and Plastic Surgery/CCT Research, Scottsdale, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - Northwest Arkansas Clinical Trials Center, PLLC, Rogers, Arkansas
  - Kern Research Inc., Bakersfield, California
  - Hope Clinical Research, Canoga Park, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - University of California, Irvine, Irvine, California
  - Dermatology Research Associates, Los Angeles, California
  - Quest Dermatology Research, Northridge, California
  - Kaiser Permanente Northern California - Oakland, Oakland, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - Stanford University School of Medicine - Medical Dermatology Clinic, Redwood City, California
  - Kaiser Permanente South Sacramento, Sacramento, California
  - Kaiser Permanente Clinical Trials Unit, San Francisco, California
  - Colorado Center for Dermatology, PLLC d/b/a CODerm Research, Centennial, Colorado
  - Colorado Medical Research Center, Denver, Colorado
  - Yale University Church Street Research Unit, New Haven, Connecticut
  - Skin Care Research, LLC, Boca Raton, Florida
  - Skin Care Research, LLC, Hollywood, Florida
  - University of Miami Hospital, Miami, Florida
  - Floridian Research Institute, LLC, Miami, Florida
  - Lenus Research & Medical Group, LLC, Sweetwater, Florida
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - ASR, LLC, Boise, Idaho
  - Denova Research, Chicago, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DS Research, New Albany, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - DS Research, Louisville, Kentucky
  - Qualmedica Research, Owensboro, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clarkston Skin Research, Clarkston, Michigan
  - Clinical Research Institute of Michigan, Clinton Township, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - University of Minnesota Department of Dermatology, Minneapolis, Minnesota
  - Vivida Dermatology, Las Vegas, Nevada
  - Skin Laser and Surgery Specialists of NJ, Hackensack, New Jersey
  - Schweiger Dermatology, P.C., Verona, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Sadick Research Group, New York, New York
  - UR Dermatology at College Town, Rochester, New York
  - Dermatology Specialists of Charlotte, Charlotte, North Carolina
  - Darst Dermatology, Charlotte, North Carolina
  - North Carolina Dermatology Associates, PLLC, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Department of Dermatology, Winston-Salem, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Remington-Davis, Inc., Columbus, Ohio
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - NW Dermatology Institute, Portland, Oregon
  - Hospital of the University of Pennsylvania Dept of Dermatology, Philadelphia, Pennsylvania
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Peak Research - Pennsylvania, Upper Saint Clair, Pennsylvania
  - Velocity Clinical Research-Providence, East Greenwich, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Palmetto Clinical Trial Services, Fountain Inn, South Carolina
  - Dermatology Treatment and Research Center - Dallas, Dallas, Texas
  - North Texas Center for Clinical Research, Frisco, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Jordan Valley Dermatology, West Jordan, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - West End Dermatology Associates, Richmond, Virginia
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin
- Canada (19):
  - Dermatology Research Institute, Calgary, Alberta
  - Kirk Barber Research, Calgary, Alberta
  - Care Clinic, Red Deer, Alberta
  - Medical Arts Health Research Group, Kelowna, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Dr. S. K. Siddha Medicine Professional Corporation, Newmarket, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - JRB research Inc., Ottawa, Ontario
  - Centre for Dermatology, Richmond Hill, Ontario
  - Research Toronto, Toronto, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain (CRDQ), Québec